CLINICAL TRIAL: NCT03960892
Title: Syrian REfuGees MeNTal HealTH Care Systems
Brief Title: Implementation of Group Problem Management Plus (PM+) in Adult Syrian Refugees in Turkey: RCT (STRENGTHS)
Acronym: (STRENGTHS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sehir University (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/2017No:2
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Anxiety; Depression; Posttraumatic Stress Disorder; Psychological Distress
Keywords: Refugees; Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-CAU with Group Problem Management Plus (PM+) (Experimental): 190 participants will be randomly assigned to E-CAU with Group PM+. The PM+ is developed by the World Health Organization (WHO) especially for the communities who are exposed to adversity. PM+ (Dawson et al., 2015) belongs to a set of programs which are low-intensity, shorter, less expensive and trans-diagnostic (i.e., not condition-specific, but targeted at a broader set of symptoms of common mental disorders) programs to reduce common mental health symptoms (including depression, anxiety and stress symptoms) and improve psychosocial functioning.
  The participants in the experimental arm will receive Group PM+ by trained, non-specialist peer-refugees in addition to E-CAU.
  Interventions: Behavioral: Problem Management Plus (PM+)
- Enhanced care as usual (E-CAU) only (No Intervention): 190 participants will be randomly assigned to E-CAU group. CAU ranges from the free health services government provides to Refugee and Asylum Seekers Assistance and Solidarity Association's (RASASA) mental health services which are provided by the Psychological Support Unit (MHPSS Support Unit) which includes counselling as well. The enhanced care arm (CAU, with the addition of a leaflet which will include information on the services that they can get from RASASA and other public services. ), is to be used as a benchmark for measuring the effectiveness of STRENGTHS's intervention, which is Problem Management Plus (PM+).

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — This intervention is based on the WHO treatment guidelines for conditions related to stress (WHO, 2013). It is a 5-session intervention that is delivered by trained non-specialists, and is available in individual and group delivery formats for both children and adults. PM+ includes evidence-based techniques such as; problem solving, stress management, behavioral activation, and accessing social support. It has proved to be effective by two randomized controlled trials (RCTs) in Kenya and Pakistan (Bryant, Dawson, Schafer, Sijbrandij, & van Ommeren, 2016; Rahman, Hamdani, Awan, Bryant, Dawson, Khan, Mukhtar-ul-Haq Azeemi, et al., 2016).
  Arms: E-CAU with Group Problem Management Plus (PM+)

SUMMARY:
To implement Group Problem Management Plus (PM+) in Syrian refugees with this RCT to evaluate feasibility, acceptability, effectiveness and cost-effectiveness of the culturally adapted Group PM+ intervention for adult Syrian refugees in Turkey.

DETAILED DESCRIPTION:
The STRENGTHS (Syrian REfuGees MeNTal HealTH Care Systems) study is a 5-year study that started in January 2017 with funding from the European Commission Horizon 2020 scheme. Turkey is one of the eight sites in STRENGTHS project that this study will be conducted. The main aim of STRENGTHS in Turkey is to evaluate the feasibility, acceptability, effectiveness and cost-effectiveness of the culturally adapted psychological intervention Group Problem Management Plus (PM+) intervention for adult Syrian refugees in Turkey.

Study participants (n=380) will consist of adult Syrian refugees (18 years and older) in Turkey with self-reported functional impairment (WHODAS 2.0 >16) and elevated psychological distress (K10 >15.9). Participants will be randomly allocated either to the treatment group who will receive five sessions of PM+ or to the enhanced care-as-usual (E-CAU) group. Participants in the comparison group will receive E-CAU only. The primary outcome will be the decrease in psychological distress from baseline to three-month post-intervention assessment, measured through the Hopkins Symptoms Checklist (HSCL-25).

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or above
* Syrian under temporary protection status
* Arabic-speaking
* Elevated levels of psychological distress (K10 >15) and reduced psychosocial functioning (WHODAS 2.0 >16)

Exclusion Criteria:

* Acute medical conditions
* Imminent suicide risk or expressed acute needs/protection risks (e.g., a young woman who expresses that she is at acute risk of being assaulted or killed)
* Severe mental disorder (psychotic disorders, substance-dependence)
* Severe cognitive impairment (e.g., severe intellectual disability or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2018-12-29 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to measure the change in psychological distress. Sub-scales can be calculated for depression (13 items) and anxiety symptoms (10 items). There are two items related to somatic symptoms. The items are rated on a 1-4 point Likert scale, with a well-validated cut-off score of 1.75. The current study will primarily look at the total score in which the lower values represent a better outcome. Furthermore, aim is to examine changes in caseness in depression, a cut-off score for the depression sub-scale of 2.1 will be used.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to measure the change in PTSD symptoms. PCL-5 is a 20-item checklist corresponding with the 20 DSM-5 PTSD symptoms. Items are rated on a 0-4 scale and add up to a total severity score of 80, with higher scores indicating worse symptomatology. The current study will primarily look at the total score in which the lower values represent a better outcome.
Psychological Outcome Measures (PSYCHLOPS) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to assess the change in self-identified problems. PSYCHLOPS consists of four questions. It contains three domains: 2 questions on problems, 1 question on function, and 1 question on well-being. Participants are asked to give free text responses to the problem and function domains. Responses are scored on a 0-5 scale producing a maximum score of 20 (six points per domain). The current study will primarily look at the total score in which the lower values represent a better outcome.
Client Service Receipt Inventory (CSRI) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to measure the change in the cost of care. CSRI was developed for the collection of data on service utilization, and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research. The current study will assess the health service utilization ad productivity impact
Access to health care: own questionnaire | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to assess the change in access to health care. The questionnaire will include 70 questions on perceived access to health care. 57 of those questions will be two-way closed ended questions (yes or no) with the addition of the items "don't know" and "refused to answer". 13 of these questions are asking the type of help received (counselling/psychotherapy, psychological support, and medicines) with the addition of the items "don't know" and "refused to answer". The current study will look at the change in the access to health care.
Socio-demographic information and disability: WHODAS | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline), and change from at 12 month post intervention assessment
  The aim is to assess the difficulties people have due to their illness across domains during the last 30 days. This questionnaire includes 12 questions scored on a five-point Likert scale ranging from 0 (none) to 4 (extreme), before summation (range 0-48). Higher scores indicate worse functional impairment.

OTHER OUTCOMES:
Traumatic experiences questionnaire: own questionnaire | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from at 12 month post intervention assessment
  The aim of the questionnaire is to assess the trauma exposure. The questionnaire has 28 items items from the Harvard Trauma Questionnaire (HTQ), and the Posttraumatic Diagnostic Scale (PDS), and specific traumatic experiences of Syrian refugees. The items scored as 1 (yes) or 0 (no), ranging from 0 to 28.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Ceren Acartürk, Assoc. Prof., Principal Investigator — Koç University
Locations (1):
- Refugee and Asylum Seekers Assistance and Solidarity Association's (RASASA), Istanbul, Sultanbeyli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The STRENGTHS project is consisted of various partners from different sites (such as the Netherlands, Jordan, Germany etc.). It is planned that the individual sites will be sharing their data with the researchers who are from these project partners. In addition to this, the partners will use the same Study Protocol while adapting it to their site.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The STRENGTHS project is a five year project which started in 2017. The individual participant data will be available for the other partners during the project which is between 2017 and 2022.
Access Criteria: The criteria for access is to be a partner of the STRENGTHS project.

REFERENCES:
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Derived] Uygun E, Ilkkursun Z, Sijbrandij M, Aker AT, Bryant R, Cuijpers P, Fuhr DC, de Graaff AM, de Jong J, McDaid D, Morina N, Park AL, Roberts B, Ventevogel P, Yurtbakan T, Acarturk C; STRENGHTS consortium. Protocol for a randomized controlled trial: peer-to-peer Group Problem Management Plus (PM+) for adult Syrian refugees in Turkey. Trials. 2020 Mar 20;21(1):283. doi: 10.1186/s13063-020-4166-x. PMID 32192539